CLINICAL TRIAL: NCT01464294
Title: Clinical Evaluation of Chairside CAD/CAM Nano-ceramic Restorations
Status: Terminated | Type: Observational
Why Stopped: not a required sutudy to be posted
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 3M ESPE CR-10-019
Record Dates: First submitted 2011-10-27; First posted 2011-11-03 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Restoration of Posterior Teeth
Keywords: CAD/CAM; crowns; onlays; composite block; milled restorations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- nano-composite: crowns and onlays
  Interventions: Device: Milled nano-composite restorations
- ceramic: crowns & onlays
  Interventions: Device: Milled ceramic restorations

INTERVENTIONS:
Device: Milled ceramic restorations — Restoration of back teeth with milled ceramic crowns or onlays
  Other Names: Empress CAD/CAM leucite porcelain (Ivoclar Vivadent)
  Groups: ceramic
Device: Milled nano-composite restorations — Restoration of back teeth with milled crowns or onlays
  Other Names: Lava Ultimate CAD/CAM Restorative (3M ESPE)
  Groups: nano-composite

SUMMARY:
Study aim is to test whether nano-composite CAD/CAM milled restorations have a similar performance in clinical service to conventional ceramic CAD/CAM restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or over
* To have at least one carious lesion or defective restoration in a molar or premolar tooth, cavities to be large enough to warrant a milled restoration of either a crown or onlay
* Teeth to be vital and asymptomatic

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth that have had root canal treatment
* Patients with significant untreated dental disease including periodontitis and rampant caries
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending and/or under clinical treatment at the University of Michigan Dental Clinics
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
clinical performance | 3 years
  Subjective evaluation of restorations using USPHS criteria

SECONDARY OUTCOMES:
Luting cement | 3 years
  Subjective evaluaton of performance of a nano-filled resin luting cement used to cement the study onlays

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fasbinder, DDS, Principal Investigator — School of Dentistry, Univ of Michigan
Locations (1):
- School of Dentistry, Unversity of Michigan, Ann Arbor, Michigan, United States